CLINICAL TRIAL: NCT03100760
Title: A Phase 1, Open-label, Evaluation of a 13C-urea Breath Test for the Detection of Urease-producing Bacteria in Patients Diagnosed With Pneumonia in the Emergency Department
Brief Title: Urease Breath Test for Rapid Characterization of Pneumonia
Status: Completed | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Avisa Pharma Inc. (Unknown); Malvern Consulting Group, Inc. (Unknown)
Responsible Party: Principal Investigator, Justin T Baca, Assistant Professor of Emergency Medicine, University of New Mexico
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 16-327
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Pneumonia, Bacterial
Keywords: urease; Point-of-Care; Breath test
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Intervention Model Description: Open label evaluation of breath test for safety and detection of urease producing pathogens in two cohorts of emergency department patients with suspected bacterial pneumonia.
Who Masked: Care Provider
Masking Description: Care Providers will not be provided with the results of the breath test, and will treat patients according to the current standards of care
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (2):
- Study of Outpatient Treatment Cohort (Experimental): Subjects presenting to the emergency department with clinical suspicion for bacterial pneumonia and plan for outpatient treatment will undergo collection of baseline breath samples (up to 6), followed by complete nebulization of 13C-urea solution. Immediately following the end of nebulization, breath collection bag samples will be collected at up to 6 time points with at least 1 minute intervals within 10 minutes post-nebulization. Exhaled breath bags will be centrally processed to determine the change in exhaled 13CO2 levels.
  Interventions: Device: 13C-urea breath test
- Study of Inpatient Treatment Cohort (Experimental): Subjects presenting to the emergency department with clinical suspicion for bacterial pneumonia and plan for inpatient treatment will undergo collection of baseline breath samples (up to 6), followed by complete nebulization of 13C-urea solution. Immediately following the end of nebulization, breath collection bag samples will be collected at up to 6 time points with at least 1 minute intervals within 10 minutes post-nebulization. Exhaled breath bags will be centrally processed to determine the change in exhaled 13CO2 levels.
  Interventions: Device: 13C-urea breath test

INTERVENTIONS:
Device: 13C-urea breath test — Subjects will undergo 13C-urea breath test involving collection of baseline breath samples, nebulization of 13C-urea, and collection of post-nebulization breath samples

SUMMARY:
This is a Phase 1, open label, evaluation of a 13C-urea breath test for the detection of urease-producing bacteria in patient with pneumonia in the emergency department.

DETAILED DESCRIPTION:
This is a Phase 1, open-label evaluation of an inhaled 13C-urea breath test in the identification of urease positive bacteria in patients diagnosed with pneumonia in the emergency department (ED). This study will enroll up to 75 adult male and female subjects in two cohorts. Adult subjects will be screened for participation in two dosing cohorts to be enrolled sequentially. Cohort A will enroll 15 subjects presenting to the ED with clinical concern for pneumonia and plan for outpatient treatment. Following enrollment and review of the safety of dosing in Cohort A, subjects receiving a diagnosis of pneumonia in the ED that are planned for admission will be screened for enrollment in Cohort B. Eligible subjects will provide informed consent, medical history, and samples for laboratory testing (including pregnancy testing for females of childbearing potential) during screening. Subjects will be evaluated for their CURB-65 Pneumonia Severity Score, and Community-Acquired Pneumonia Severity Index (PSI) where required data are available.

Prior to breath test administration, subjects will provide a sputum sample for bacterial culture; sample may be induced, or collected as part of initial ED workup if appropriate culture has been ordered. Subjects will undergo breath test with collection of baseline breath samples (up to 6), followed by complete nebulization of 13C-urea solution. Immediately following the end of nebulization, breath collection bag samples will be collected at up to 6 time points with at least 1 minute intervals within 10 minutes post-nebulization. Exhaled breath bags will be centrally processed to determine the change in exhaled 13CO2 levels. Vital signs, including resting blood pressure, resting pulse, respiratory rate, peripheral oxygen saturation, and temperature will be collected prior to, and following completion of, nebulization treatment. In the event of bronchospasm, during or following nebulization, albuterol rescue will be available for treatment at the discretion of the investigator.

Once required tests are complete, the subject will be treated/followed according to standard institutional protocol/practice. The subjects' clinical course will be followed for at least 24 hours, where possible, to document the final diagnosis and outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort A Only: be a man or woman age 18-65, inclusive, with suspected bacterial pneumonia on presentation to the ED based on clinical signs and symptoms AND be planned for outpatient treatment

   OR

   Cohort B Only: be a man or woman age 18-85, inclusive, with a diagnosis of suspected bacterial pneumonia in the ED based on findings of a positive chest x-ray and clinical signs and symptoms AND be planned for admission to the hospital ward/floor
2. be capable of providing a spontaneous or induced sputum sample for analysis
3. be capable of completing the breath test according to the clinical judgement of the investigator
4. be able to understand the study procedures, agree to participate in the study program, and voluntarily provide written informed consent

Exclusion Criteria:

1. have a known allergy to urea or any excipient in the nebulized solution
2. be pregnant or have a positive urine pregnancy test
3. have evidence of active oral infection, such as abscess or dense exudate, that requires antibiotic therapy
4. have known diagnosis of cystic fibrosis or bronchiectasis
5. have a known or suspected acute asthma exacerbation on presentation to the ED
6. have received treatment with oral or intravenous (IV) antibiotics in the preceding 2 days prior to screening, unless antibiotic failure is suspected

   OR

   have received treatment in the ED with oral or IV antibiotics greater than 4 hours prior to breath test
7. have an acute illness or other condition that, as determined by the investigator, would preclude participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the emergency departments of University of New Mexico Health Sciences Center and Henry Ford Hospital. Eligible participants presented with clinical suspicion for community-acquired pneumonia and were screened for outpatient (Cohort A) or inpatient (Cohort B) treatment enrollment.
Pre-assignment Details: All subjects provided written informed consent prior to participation. Subjects were screened for eligibility, including medical history, vital signs, and ability to perform breath sampling. No randomization was performed; subjects were assigned to outpatient or inpatient cohorts based on clinical treatment plan.
Groups:
- Outpatient Treatment Cohort (Cohort A): Subjects with suspected bacterial pneumonia planned for outpatient treatment who received the 13C-urea breath test.
- Inpatient Treatment Cohort (Cohort B): Subjects with suspected bacterial pneumonia planned for inpatient hospital admission who received the 13C-urea breath test.
Period: Overall Study
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Started | 15 | 60
Completed | 15 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who enrolled and completed breath testing are included in the baseline analysis population. No exclusions were made. Participant totals reflect completion at both study sites.
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B) | Total
Number analyzed (Participants) | 15 | 60 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years at time of study enrollment.
  Years | 45 (14) | 60 (14.6) | 54 (14)
Sex: Female, Male [Count of Participants; unit: Participants] — Number and percentage of participants who self-identified as female or male at enrollment.
  Participants
    Female | 9 | 28 | 37
    Male | 6 | 32 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data were collected for inpatient participants but not outpatient participants. Population: Race data were collected for inpatient participants but not outpatient participants.
  Participants
    number analyzed (Participants) | 0 | 60 | 60
    American Indian or Alaska Native | 0 | 5 | 5
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 0 | 15 | 15
    White | 0 | 34 | 34
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity data were collected for inpatient participants but not outpatient participants. Population: Ethnicity data were collected for inpatient participants but not outpatient participants.
  Participants
    number analyzed (Participants) | 0 | 60 | 60
    Hispanic or Latino | 0 | 15 | 15
    Not Hispanic or Latino | 0 | 42 | 42
    Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled at U.S. clinical sites (University of New Mexico Health Sciences Center and Henry Ford Hospital).
  Participants
    United States | 15 | 60 | 75

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Time Frame: Within 24-48 hours of breath test
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 15 | 60
Participants
  Brief Coughing | 3 | 0
  Nausea | 1 | 0
  Syncope 24 hours post nebulization | 1 | 0

2. Primary Outcome: Serious Adverse Events
Description: Death, disability, incapacitation, escalation of level of care, prolongation of hospitalization, birth defect, or intervention to prevent the above.
Time Frame: Within 24-48 hours of breath test
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 15 | 60
Participants | 0 | 0

3. Primary Outcome: Suspected Adverse Reaction
Description: Any adverse event for which there is a reasonable possibility that the adverse event was caused by the study drug.
Time Frame: Within 24-48 hours of breath test
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 15 | 60
Participants | 0 | 0

4. Primary Outcome: Serious Suspected Adverse Reaction
Description: Any Suspected Adverse Reaction that is determined to be serious, based on the outcomes of a Serious Adverse Event; i.e. death, life-threatening, causes or prolongs inpatient hospitalization, causes a persistent of significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital abnormality/birth defect.
Time Frame: Within 24-48 hours of breath test
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 15 | 60
Participants | 0 | 0

5. Secondary Outcome: Exhaled 13CO2 Concentration
Description: We recorded change in 13CO2/12CO2 ratio (delta over baseline or ΔOB, in units of ‰) between pre- and post-nebulization samples
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Population: We recorded change in 13CO2/12CO2 ratio (delta over baseline or ΔOB, in units of ‰) between pre- and post-nebulization samples
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 15 | 60
Percent change | 1.3 (1.2) | 14.92 (30.26)

6. Secondary Outcome: Number of Participants With ¹³CO₂/¹²CO₂ Ratio Correlated (ρ > 0.75) to Bacterial RNAseq Counts
Description: We recorded change in 13CO2/12CO2 ratio (delta over baseline or ΔOB, in units of ‰) between pre- and post-nebulization samples and compared with subject's causative pathogen based upon sputum or blood culture results
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Population: The change in 13CO2/12CO2 ratio (delta over baseline or ΔOB, in units of ‰) between pre- and post-nebulization samples was compared to RNAseq bacterial counts. Positive relationships and/or correlations were tested using Spearman's rank correlations. A Spearman value above 0.75 was selected as the cutoff, above which results would be determined to be a positive outcome. A spearman correlation > 0.75 for any bacteria, the subject would be a positive outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 8 | 30
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With ¹³CO₂/¹²CO₂ Ratio Correlated (ρ > 0.75) to CURB-65 Score in Urease-Positive Pneumonia
Description: Number of participants With ¹³CO₂/¹²CO₂ Ratio Correlated (ρ > 0.75) to CURB-65 Score in Urease-Positive Pneumonia
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Population: Linear regression and Spearman correlation was used to determine if CURB65 score correlated with the change in 13CO2 divided by the baseline 13CO2. A spearman correlation > 0.75 and/or a coefficient of determination > .70 would mean the subject was listed as a positive outcome in the data table.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 8 | 30
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With ¹³CO₂/¹²CO₂ Ratio Correlated (ρ > 0.75) to Pneumonia Severity Index in Urease-Positive Pneumonia.
Description: Number of Participants With ¹³CO₂/¹²CO₂ Ratio Correlated (ρ > 0.75) to Pneumonia Severity Index in Urease-Positive Pneumonia.
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 8 | 30
Participants | 0 | 0

9. Secondary Outcome: Number of Participants Meeting Sensitivity Criterion of ¹³C-Urea Breath Test for Urease-Producing Pathogens
Description: This exploratory outcome was designed to assess whether the ¹³C-urea breath test (Δ¹³CO₂) is associated with the presence of urease-producing pathogens. Correlation between exhaled ¹³CO₂ levels and pathogen abundance (based on RNAseq bacterial counts) was to be evaluated using Spearman's correlation, with a pre-defined significance threshold of ρ > 0.75.
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Population: Participants with both breath test data and RNAseq-based bacterial abundance profiles were included in this analysis. Urease-producing pathogens were identified based on taxonomy and literature-reported activity. The outcome was defined as the number of participants with a Spearman correlation coefficient greater than 0.75 between Δ¹³CO₂ and pathogen abundance.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 8 | 30
Participants | 0 | 0

10. Secondary Outcome: Number of Participants Meeting Specificity Criterion of ¹³C-Urea Breath Test for Urease-Producing Pathogens
Description: This exploratory outcome was designed to assess the specificity of the ¹³C-urea breath test (Δ¹³CO₂) for detecting urease-producing pathogens. Specificity was defined as the proportion of participants without urease-producing pathogens (based on RNAseq bacterial profiles) who also did not meet the predefined breath test threshold. The planned analysis used Spearman correlation (ρ) between ¹³CO₂ enrichment and bacterial abundance, with ρ < 0.75 indicating a negative test result.
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Population: Participants without RNAseq-detected urease-producing pathogens and with available breath test data were included in this analysis. A specific breath test response was defined as Spearman ρ > 0.75 between Δ¹³CO₂ and pathogen abundance. Participants not meeting this criterion were considered test-negative. The outcome measured the proportion of participants correctly classified as negative by the breath test.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 8 | 30
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Breath Test Positive and Confirmed Urease-Producing Pathogen (PPV Criterion)
Description: This exploratory outcome measured the number of participants who met the criteria for positive predictive value of the ¹³C-urea breath test. A participant was considered to meet the PPV criterion if they had a positive breath test result (Spearman ρ > 0.75 between Δ¹³CO₂ and bacterial abundance) and also had RNAseq-confirmed presence of at least one urease-producing pathogen.
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Population: Participants with both ¹³C-urea breath test results and RNAseq bacterial profiling were included in this analysis. Positive breath test results were defined by Spearman correlation ρ > 0.75 between Δ¹³CO₂ and bacterial abundance. Urease-producing pathogens were identified based on taxonomic classification and known enzymatic activity. The outcome was the count of participants meeting both conditions.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 8 | 30
Participants | 0 | 0

12. Secondary Outcome: Number of Participants Meeting Negative Predictive Value Criterion of ¹³C-Urea Breath Test for Urease-Producing Pathogens
Description: This exploratory outcome was designed to evaluate the number of participants meeting the negative predictive value (NPV) criterion of the ¹³C-urea breath test for detecting urease-producing pathogens. A participant was considered to meet the NPV criterion if they had a negative breath test result defined as a Spearman correlation coefficient (ρ) ≤ 0.75 between Δ¹³CO₂ and bacterial abundance and RNAseq-confirmed absence of urease-producing pathogens.
Time Frame: Collected at 6 minutes after nebulization and measured within 7 days of collection
Population: Participants with both ¹³C-urea breath test data and RNAseq bacterial profiles were included in this analysis. Breath test negativity was pre-defined as Spearman ρ ≤ 0.75. Participants without detectable urease-producing pathogens based on RNAseq taxonomic analysis were considered pathogen-negative. The outcome represents the number of participants who were both test-negative and pathogen-negative.
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
Number analyzed (Participants) | 8 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From immediately after 13C-urea breath test to 24-48 hours post-dose
Arm/Group | Outpatient Treatment Cohort (Cohort A) | Inpatient Treatment Cohort (Cohort B)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/60
Other Adverse Events (participants affected / at risk) | 5/15 | 0/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Treatment Cohort (Cohort A) (N=15) | Inpatient Treatment Cohort (Cohort B) (N=60)
Coughing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — brief coughing, which resolved spontaneously
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — nausea, which was mild and self-limited
Syncope (Cardiac disorders) | 1 (1) | 0 (0) — syncope occurred 24 hours after nebulization

LIMITATIONS AND CAVEATS:
Small sample size, observational design, and limited follow-up period may limit generalizability. Study was primarily designed to assess safety and feasibility, not diagnostic efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03100760/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort B (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT03100760/ICF_001.pdf
  • Informed Consent Form: Cohort A (2017-08-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT03100760/ICF_002.pdf